CLINICAL TRIAL: NCT01474863
Title: Prospective, Randomized, Double-Blind, Placebo-Controlled Phase II Trial of Intravenous Citrulline to Prevent or Mitigate Acute Lung Injury in Patients With Severe Sepsis
Brief Title: Citrulline in Severe Sepsis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Todd Rice, Assistant Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 111435
Record Dates: First submitted 2011-11-11; First posted 2011-11-18 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Severe Sepsis; Acute Lung Injury
MeSH Terms: conditions — Sepsis; Acute Lung Injury | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose Citrulline (Active Comparator): Low Dose Citrulline
  Interventions: Drug: Low Dose Citrulline
- Placebo (Placebo Comparator): Placebo IV infusion
  Interventions: Drug: Placebo
- High Dose Citrulline (Active Comparator): High Dose Citrulline
  Interventions: Drug: High Dose Citrulline

INTERVENTIONS:
Drug: High Dose Citrulline — Initial intravenous bolus of 20mg/kg (to a maximum of 1500mg) L-citrulline over 10 minutes. Immediately after the initial bolus, a continuous intravenous infusion of L-citrulline at 9mg/kg (max 700mg) per hour will be administered through a dedicated intravenous line or port of a multilumen catheter for 4 days
  Arms: High Dose Citrulline
Drug: Placebo — D5W IV fluids at isovolumetric rate (about 15ml/hr)
  Arms: Placebo
Drug: Low Dose Citrulline — Initial intravenous bolus of 10mg/kg (to a maximum of 1500mg) L-citrulline over 10 minutes. Immediately after the initial bolus, a continuous intravenous infusion of L-citrulline at 4.5mg/kg (max 350mg) per hour will be administered through a dedicated intravenous line or port of a multilumen catheter for 4 days.
  Arms: Low Dose Citrulline

SUMMARY:
This is a randomized, double-blind, placebo-controlled, phase 2 study to evaluate biochemical, clinical, and safety effects of 2 doses of intravenous L-citrulline compared to placebo in patients with severe sepsis at risk for or with acute lung injury. The hypothesis is that intravenous L-citrulline will decreased the development or progression of acute lung injury in patients with severe sepsis compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Severe Sepsis

Exclusion Criteria:

* No Consent
* Malignant or other irreversible condition
* Moribund and not expected to survive 48 hours
* End Stage Liver Disease
* Enrolled in another IND study
* Pregnant or breast feeding female
* Age<13 years old
* Allergy to citrulline or arginine

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Rice, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose Citrulline | Placebo | High Dose Citrulline
Started | 26 | 22 | 24
Completed | 26 | 22 | 24
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Citrulline | Placebo | High Dose Citrulline | Total
Number analyzed (Participants) | 26 | 22 | 24 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (17.1) | 56.2 (16.8) | 51.8 (16.6) | 54.1 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 12 | 30
  Male | 16 | 14 | 12 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 2 | 9
  White | 23 | 18 | 22 | 63
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 22 | 24 | 72

OUTCOME MEASURES:

1. Primary Outcome: Vasopressor Dependency Index
Description: Worst Value of Index measuring blood pressure hourly through study infusion (day 4). Vasopressor index is mean arterial blood pressure divided by catecholamine index (the catecholamine index is a dimensionless variable calculated as (dopamine dose × 1) + (dobutamine dose × 1) + (adrenaline dose × 10) + (noradrenaline × 100) + (phenylephrine dose × 100), where all doses are expressed in ug/kg/min). (Higher is better)
Time Frame: day 4
Measure: Mean (Standard Deviation); unit: mmHg/catecholamine index
Arm/Group | Low Dose Citrulline | Placebo | High Dose Citrulline
Number analyzed (Participants) | 26 | 22 | 24
mmHg/catecholamine index | 50.0 (28.8) | 44.4 (30.9) | 49.0 (27.4)
Statistical Analysis 1: Comparison: Low Dose Citrulline vs Placebo vs High Dose Citrulline; Test type: Superiority; p = 0.86, ANOVA

ADVERSE EVENTS:
Arm/Group | Low Dose Citrulline | Placebo | High Dose Citrulline
All-Cause Mortality (participants affected / at risk) | 5/26 | 5/22 | 3/24
Serious Adverse Events (participants affected / at risk) | 5/26 | 5/22 | 3/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/22 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Citrulline (N=26) | Placebo (N=22) | High Dose Citrulline (N=24)
Death (Cardiac disorders) | 5 (5) | 5 (5) | 3 (3) — Death

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No